CLINICAL TRIAL: NCT02800668
Title: Metabolic Effects of Duodenal Jejunal Bypass Liner for the Treatment of Adipose Patients With Type 2 Diabetes Mellitus
Brief Title: Metabolic Effects of Duodenal Jejunal Bypass Liner for Type 2 Diabetes Mellitus
Acronym: DJBL-T2DM
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Diethelm Tschoepe, Prof. Dr. Dr., Ruhr University of Bochum
Other Study IDs: DJBL-HDZ
Record Dates: First submitted 2016-05-25; First posted 2016-06-15 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
Keywords: Duodenal Jejunal Bypass Liner; obesity; weight loss therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood sampling during study, analysis via ELISA for special markers at study end in one batch, active medical control parameters like HbA1c, cholesterol, hemogram etc. at visits
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DJBL implant-group: T2DM Patients implanted with a DJBL (Duodenal jejunal Bypass liner, EndoBarrier, GI Dynamics) due to medical reasons.
  The subjects were regular in-patients of the Diabetes Center at the Heart and Diabetes Center NRW, Germany and gave informed consent for related procedures and data handling. The subjects had BMI ≥35 kg/m2, T2DM, and a history of frustrated weight loss attempts. Exclusion criteria: history of gastric surgery, gastric or duodenal ulcers, thyroid disorders, gastrointestinal disorders with intestinal resorption dysfunction, therapy with oral anticoagulants, use of acetyl salicylic acid or non-steroidal anti-inflammatory drugs, drug abuse (incl. alcohol), symptomatic cardiovascular disease, renal insufficiency (GFR <50 ml/min), pregnancy or breast feeding.
  Interventions: Device: DJBL (Duodenal jejunal bypass liner, EndoBarrier)

INTERVENTIONS:
Device: DJBL (Duodenal jejunal bypass liner, EndoBarrier) — Implantation of EndoBarrier after medical and patient's decision, Duration of treatment 12 months in maximum, follow up for 4 weeks after Explantation, follow up during treatment by physical examination, ECG control, sampling and analysis of blood parameters, mixed meal tolerance tests only for diagnostic purposes to assess gut hormonal changes and metabolic parameters
  Other Names: EndoBarrier

SUMMARY:
Implantation of a duodenal-jejunal endoluminal bypass liner (DJBL) has shown to induce weight loss and to improve metabolic parameters. DJBL is a reversible endoduodenal sleeve mimicking biliodigestive digestion while lacking risks and limitations of bariatric surgery.

Effects on metabolic control, body mass parameters, appetite regulation, glucose tolerance, organ health, and lipid profile were determined in 16 morbidly overweight patients with type 2 diabetes mellitus. In addition, relevant hormones (Leptin, ghrelin, gastric inhibitory peptide, glucagon-like peptide 1, and insulin) were measured by enzyme-linked immunosorbent assay (ELISA) and chemiluminescent microparticle immunoassay (CMIA) at 0, 1 and 32, and 52 weeks post-implant following a mixed meal tolerance test, which was applied for diagnostic purposes only.

DETAILED DESCRIPTION:
A total of 18 subjects (4 women and 14 men) aged 39 to 66 years underwent implantation of the DJBL.The subjects were regular patients of the Diabetes Center at the Herz- und Diabeteszentrum Nordrhein-Westfalen (HDZ NRW), Germany and gave informed consent for related procedures and data handling. The subjects had body mass index (BMI) ≥35 kg/m2, type 2 diabetes mellitus (T2DM), and a history of frustrated weight loss attempts. Exclusion criteria were: history of gastric surgery, gastric or duodenal ulcers, thyroid disorders, gastrointestinal disorders associated with intestinal resorption dysfunction, therapy with oral anticoagulants like marcumar, use of acetyl salicylic acid or non-steroidal anti-inflammatory drugs, drug abuse (incl. alcohol), symptomatic cardiovascular disease including heart failure New York Heart Association (NYHA) IV, renal insufficiency defined as glomerular filtration rate (GFR) <50 ml/min, pregnancy or breast feeding.

Study design All patients received the DJBL due to medical reasons, not for study purposes. All patients underwent pre-implantation and follow-up examinations (1 week, 32 weeks and 52 (explantation) weeks after implantation). Every examination included a thorough body examination, electrocardiogram (ECG), and the body composition measurement by bio-impedance scaling (type: BC418MA, Tanita, Amsterdam, the Netherlands). Upon implantation, antidiabetic medication was adapted, patients were followed up to adjust antidiabetic regimen. Dietary advice was given to the patients by a professional dietician upon implantation procedure, and liquid diet was started the day before implantation and continued for two additional days followed by puréed diet for four days. Patients decided to turn back to normal diet upon tolerance; fibre rich dietary components were prohibited during the treatment period. Treatment with glucagon-like peptide-1 (GLP-1) or dipeptidyl-peptidase-4 (DPP4) based medication (Exenatide, Liraglutide, Lixisenatide or Sitagliptin, Vildagliptin) was initiated in cases that fasting C-peptide levels were >750 pmol/l. Insulin dosage was reduced after implantation to avoid risk of hypoglycaemia. Sulfonylurea treatment was stopped after implantation.

Mixed meal tolerance tests Mixed meal tolerance tests (MMTT) were performed in fasting state as routine diagnostic tool to assess metabolism parameters and gut hormones described below. In the course of a MMTT every patient consumed a highly caloric drink (Fortimel regular 2 093 Kilojoules (KJ), Nutricia GmbH, Erlangen, Germany) containing carbohydrates (41 energy(EN)%), proteins (40 EN%) and fats (19 EN%), simulating an average meal. Blood samples were taken at fixed intervals: before drinking, after 10, 30, 60, 90, 120 min. DPP4 inhibitor was added to prevent autodigestion of GLP-1 immediately after sampling, Hydroxymercuribenzoic acid was added to plasma per protocol to prevent ghrelin digestion. Samples were stored after centrifugation at -80°C until assayed for the gut hormones ghrelin, GLP-1, gastric inhibitory peptide, leptin as well as the metabolism parameters glucose, insulin, C-peptide, and proinsulin.

Biochemical assessment Laboratory assessments were done in fasting state. Venipuncture was performed the morning after overnight fasting one day before the planned procedure, one week, 8, and 12 months after implantation. Blood samples were processed for subsequent analysis within 20 min of venipuncture. Serum concentrations were measured by commercial available kits of total ghrelin (ELISA, Merck Chemicals Gesellschaft mit beschränkter Haftung (GmbH), Schwalbach, Germany), leptin (ELISA, DRG-International, Inc., USA), active GLP-1 (ELISA, epitope Diagnostics, San Diego, USA), gastric inhibitory Peptide (GIP) (ELISA, DRG-International, Inc., USA), Insulin (CMIA, Abbott, Wiesbaden, Germany), C-peptide (CMIA, Abbott, Wiesbaden, Germany), Proinsulin (ELISA, TecoMedical Bunde, Germany) and glucose (CMIA, Abbott, Wiesbaden Germany).

ELIGIBILITY:
Inclusion Criteria:

* T2DM
* body mass index (BMI) ≥35 kg/m2
* history of frustrated weight loss attempts

Exclusion Criteria:

* history of gastric surgery, gastric or duodenal ulcers
* thyroid disorders
* gastrointestinal disorders associated with intestinal resorption dysfunction
* therapy with oral anticoagulants like marcumar
* use of acetyl salicylic acid or non-steroidal anti-inflammatory drugs
* drug abuse (incl. alcohol)
* symptomatic cardiovascular disease including heart failure New York Heart Association IV
* renal insufficiency defined as GFR <50 ml/min
* pregnancy or breast feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects were regular inpatients with type 2 Diabetes mellitus of the Diabetes Center at the Heart and Diabetes Center NRW, Germany and gave informed consent for related procedures and data handling
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2011-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
weight loss in kg | 12 months
  weight loss defined as excess weight loss

SECONDARY OUTCOMES:
Change in body fat in %, measured via bioimpedance scaling | 12 months
  effect of DJBL on body composition in overweight T2DM patients determined by bioimpedance scaling
Change in HbA1c in mmol/mol | 12 months
  effect of DJBL on metabolic regulation in overweight T2DM patients
Change in LDL-cholesterol in mg/dl | 12 months
  effect of DJBL on metabolic regulation in overweight T2DM patients
Change in triglycerides in mg/dl | 12 months
  effect of DJBL on metabolic regulation in overweight T2DM patients
Change in liver enzyme aspartate aminotransferase (ASAT) in U/l | 12 months
  effect of DJBL on metabolic regulation in overweight T2DM patients
Change in liver enzyme alanine aminotransferase (ALAT) in U/l | 12 months
  effect of DJBL on metabolic regulation in overweight T2DM patients
changes in intestinal enzyme levels (GLP-1) in pmol/l/120 min during mixed meal tolerance test | 12 months
  effect of DJBL and intestine/pancreatic axis for metabolic control
changes in intestinal enzyme levels (GIP) in ng/ml/120 min during mixed meal tolerance test | 12 months
  effect of DJBL and intestine/pancreatic axis for metabolic control
changes in Ghrelin in ng/ml/120 min during mixed meal tolerance test | 12 months
  effect of DJBL and intestine/pancreatic axis for metabolic control
changes in Leptin in ng/ml/120 min during mixed meal tolerance test | 12 months
  effect of DJBL and intestine/pancreatic axis for metabolic control
changes in pancreatic enzyme levels (Insulin) in U/l/120 min during mixed meal tolerance test | 12 months
  effect of DJBL and intestine/pancreatic axis for metabolic control
changes in pancreatic enzyme levels (Proinsulin) in nmol/l/120 min during mixed meal tolerance test | 12 months
  effect of DJBL and intestine/pancreatic axis for metabolic control
effect on blood pressure measured in mmHg | 12 months
  follow up by regular vital signs,

CONTACTS AND LOCATIONS:
Overall Officials: Diethelm Tschoepe, Prof MD, Principal Investigator — Herz und Diabeteszentrum NRW
Locations (1):
- Herz- und Diabeteszentrum, Bad Oeynhausen, Germany

IPD SHARING:
Plan to Share IPD: Yes
after publication of results